CLINICAL TRIAL: NCT06088498
Title: Augmented Reality as an Adjunct to Quitline Counseling for Smoking Cessation
Brief Title: App for Reducing Cravings to Smoke
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MCC-21980 Aim 2; R01DA055298 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aim 1: Update an existing smartphone App (Experimental): An existing study app will be updated to be engaging, user-friendly treatment tool, and verify user satisfaction.
  Interventions: Behavioral: Quitline Services and Smartphone App
- Aim 2: Quit Line Only (Experimental): Participants randomized to this arm will receive usual care for smoking cessation via the quitline and a smartphone app that will allow them to track smoking urges and abstinence.
  Interventions: Behavioral: Quitline Services
- Aim 2:Quitline plus smartphone App (Experimental): Participants randomized to this arm will receive usual care for smoking cessation via the quitline and a smartphone app that will allow them to track smoking urges and abstinence. After 48 hours of self-reported abstinence, they will be exposed to smoking extinction trials through the study smartphone app.
  Interventions: Behavioral: Updating Existing Smartphone App; Behavioral: Quitline Services; Behavioral: Quitline Services and Smartphone App

INTERVENTIONS:
Behavioral: Updating Existing Smartphone App — Participants will be asked to use a recently developed study smartphone application to reduce cravings to smoke for a 5-week period. Through the app, participants will be exposed to smoking extinction trials daily. Participants will be encouraged and reminded to complete 2-5 extinction sessions per day. Each session will present 3-8 cues, and each cue will be presented for 20-40 seconds (average amount of extinction per day will be about 10 minutes). Participants will be encouraged to conduct the extinction sessions when high cravings are expected.
  Arms: Aim 2:Quitline plus smartphone App
Behavioral: Quitline Services — Quitline coaches use cognitive behavioral therapy, reinforcement, and principles of self-efficacy to promote effective behavior change. The quitline approach includes 5 key elements: setting a quit date, coping with triggers, effectively using medications, tobacco proofing, and social support. Individuals who enroll in the quitline's multi-call program receive phone calls and NRT.
  Arms: Aim 2: Quit Line Only; Aim 2:Quitline plus smartphone App
Behavioral: Quitline Services and Smartphone App — In addition to quitline services, participants will download a study app that will allow them to track smoking urges and abstinence. After 48 hours of self-reported abstinence, those in the intervention group will be exposed to smoking extinction trials through the study smartphone app.
  Arms: Aim 1: Update an existing smartphone App; Aim 2:Quitline plus smartphone App

SUMMARY:
The overall goal of the study is to assess the efficacy of using cue exposure delivered via a smartphone application as an adjunct to Tobacco Quitline treatment to improve smoking abstinence.

DETAILED DESCRIPTION:
The aims of the study are: (1) to update a recently developed study-related smartphone application to reduce cravings to smoke to be an engaging, user-friendly treatment tool, and verify user satisfaction; and (2) to test in a randomized controlled trial the efficacy of the app as an adjunct to quitline smoking cessation treatment in improving smoking abstinence compared to the quitline only.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Daily smokers that have quit smoking within the past 3 months (Aim 1) or currently smoking ≥ 3 cigarettes per day for the past year (Aim 2)
* Functioning telephone number
* Owns a smart phone capable of supporting AR and willing to download the app
* Can speak, read and write in English

Exclusion Criteria:

* Has another household member already enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (Aim 1) | At 1 Week
  Participants' perception of usability and learnability of the app will be measured using 10 items on a 5-point Likert scale. Scores range from 0 to 100, with higher scores indicating better usability.
Tobacco Abstinence (Aim 2) | At 6 Months
  Self-report of no combustible tobacco use in the past 7 days

SECONDARY OUTCOMES:
User Satisfaction (Aim 1) | At 1 Week
  One Likert scale item will capture participants' satisfaction with the app. The Likert scale is from 1 to 4, with higher score indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Vinci, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Poudel R, Dougan SO, Yates H, Sawyer L, Martinez U, Brandon KO, Sutton SK, Vidrine DJ, Ritterband LM, Wiseman KP, Vickerman KA, Turner K, Byrne MM, Yang MJ, Horta M, Brandon TH, Vinci C. Using augmented reality to deliver cue exposure treatment for smoking cessation: App usability findings and protocol for a randomized controlled trial. Contemp Clin Trials. 2025 Mar;150:107827. doi: 10.1016/j.cct.2025.107827. Epub 2025 Jan 27. PMID 39880329
- See also: Moffitt Cancer Center Clinical Trial Search — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE